CLINICAL TRIAL: NCT06650410
Title: Virtual Intervention for Vertebral frActure: a Pilot, Feasibility Study for a Multicentre Randomized Controlled Trial
Acronym: VIVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Unity Health (Other); Arthritis Research Centre of Canada (Other); Hamilton Health Sciences Corporation (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4816
Record Dates: First submitted 2024-09-25; First posted 2024-10-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis; Fractures, Spinal
Keywords: Rehabilitation; Spine fracture; Exercise; Physical functioning
MeSH Terms: conditions — Osteoporosis; Spinal Fractures; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to one of two arms. The study includes a wait-list control, indicating all participants will receive the intervention but at different time points. One group will receive the intervention immediately, whereas the other group will receive the intervention 10 weeks after being randomized (wait-list control).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be blind to group allocation of participants. Participants will not be blind to group allocation because they will know what group they are assigned to. The randomization sequence will be created and maintained using REDCap and will be conducted by exercise professionals delivering the intervention who are not blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate receipt group (Experimental): Participants in this group will receive the VIVA intervention in the first 8 weeks of the study. After the 8-week period, participants will be asked to practice behaviour change techniques for the next 10 weeks.
  Interventions: Other: Virtual Intervention for Vertebral Fractures (VIVA)
- Wait-list control and delayed receipt group (Other): Participants in this group will continue with their usual care for the first 10 weeks of the study. At week 10, they will receive the same VIVA intervention.
  Interventions: Other: Virtual Intervention for Vertebral Fractures (VIVA)

INTERVENTIONS:
Other: Virtual Intervention for Vertebral Fractures (VIVA) — VIVA is an intervention for people with vertebral fractures that covers four areas: pain management, safe movement, exercise, and nutrition. It includes print and video resources, and a framework for goal setting, selecting exercises, and teaching body mechanics. An exercise professional leads 1:1 once-weekly sessions (in person or virtual) over eight weeks. Sessions start with brief education on a topic, followed by training and modeling of exercise and safe movement strategies, then goal setting, and action planning. The exercise professional prescribes resources using an app or that can be emailed or mailed. Exercises are tailored to the participant's abilities, and target balance, muscle strength, and endurance of back extensor muscles and scapular stabilizers.

SUMMARY:
Spine fractures are the most common fracture due to osteoporosis. They happen during falls or activities of daily life, like bending to tie shoes. Fractures of the spine can result in pain, which can sometimes last for a long time. Spine fractures can affect breathing, appetite, digestion, and mobility, and can restrict or modify people's work or daily activities. There are no standard rehabilitation programs after spine fracture, and patients often have to pay for rehabilitation. Rehabilitation can be hard to access, especially in rural or remote locations. It can be hard to find health care or rehabilitation providers who specialize in treating spine fractures. After reviewing research and consulting patients and health care providers to understand their experiences with spine fracture rehabilitation, the research team developed a toolkit for a virtual rehabilitation program for people with spine fractures, called VIVA.

The research team wants to submit a grant for a clinical trial to implement VIVA in five provinces and determine if VIVA reduces pain and improves physical functioning and quality of life, and if the benefits outweigh the costs. Before this, the team proposes to do a pilot study to test how feasible it is to do a study of VIVA in three provinces.

DETAILED DESCRIPTION:
A multicenter trial will be conducted to investigate the feasibility of a future trial of VIVA in adults with spine fractures in Ontario, British Columbia, and Quebec. As secondary outcomes, the research team will explore the effect of the intervention on physical function and balance, pain, fear of movement, falls, falls self-efficacy, quality of life, mood, nutrition risk, and physical activity. Adults over the age of 50 who have had at least one spine fracture in the past two years due to osteoporosis will be recruited. Participants will be randomized either to the immediate receipt of VIVA intervention; or delayed receipt of VIVA 10 weeks post-randomization. The VIVA intervention involves once weekly 1:1 rehabilitation sessions delivered by an exercise professional for eight weeks. The study will take place at the GERAS Centre (Ontario), Unity Health (Ontario), University of British Columbia (British Columbia), and McGill University Health Centre (Quebec). University of Waterloo will be the coordinating centre. The findings of this study will be used to decide if a larger clinical trial is feasible.

ELIGIBILITY:
Inclusion Criteria:

* have had at least one vertebral fracture in the past two years confirmed by a radiology report
* willing to participate in once weekly virtual rehabilitation sessions for 8 weeks
* have access to internet and a smart device with a camera and microphone.

Exclusion Criteria:

* have cauda equina syndrome or spinal cord injury or spinal cord injury
* had a traumatic fracture (i.e., car accident); an active infection; active inflammatory arthritis with a flare up within the past two years
* an inability to follow two-step commands or understand instructions and are without a caregiver to support participation
* been participating in a similar rehabilitation program for vertebral fractures delivered by a physical therapist, exercise physiologist or kinesiologist and includes exercise
* any surgeries planned or health problems that might cause their health to change significantly in the next 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Adherence | Through the 8-week intervention period
  The adherence will be reported as the proportion of scheduled sessions participants attend.
  A future trial will be feasible if the adherence to the intervention sessions is 75%.
Recruitment | Through the 5-month recruitment period
  The recruitment will be reported as the number of participants recruited by each site.
  Feasibility criteria for recruitment will be satisfied if we recruit 8 people per site in five months.
Retention | Through study completion (18 weeks)
  The retention will be reported as the proportion of participants who complete the final assessment out of the total number of participants.
  The feasibility criteria for retention will be satisfied if 80% of participants complete the trial.

SECONDARY OUTCOMES:
Resource use | Baseline, Week 9, and Week 18
  The economic evaluation will be conducted from health system and societal perspectives using questionnaires. Participants will complete EQ5D-3L as a measure of morbidity and multiply it by mortality to achieve a quality-adjusted life year (QALY) estimate per intervention. Multiplying resources collected by jurisdictional unit costs in Canadian dollars will determine the total cost. The ratio of incremental costs between arms will be calculated, determined by trial resources, and outcome (QALY) to achieve a cost per life year gained outcome.
Implementation | At Week 18
  The participant and provider experiences will be captured via semi-structured interviews. Participants will report adherence to the prescribed exercise using Wibbi app or a log (participant preference). With consent, two sessions per site, selected at random, will be recorded. Research assistant will complete a checklist to assess intervention fidelity.
Pain level | Baseline, Week 9, and Week 18
  Participants will be administered the Brief Pain Inventory Short Form to assess pain. The wording of the questions will be modified to adapt them to the context specific to our population. The mean score of the four items will be calculated to determine pain severity, ranging from 0 to 10. The pain interference will be calculated as the mean score of 10 items that measure the impact of pain on various activities, ranging from 0 to 10.
Falls self-efficacy | Baseline, Week 9, and Week 18
  Participants will complete Short Falls Self-Efficacy questionnaire to assess fear of falling. The cut-points for degrees of concern about falling are established wherein scores 7 and 8 represent a low concern, 9 to 13 indicate a moderate concern, and 28 to 64 represent a high concern for falls.
Mood | Baseline, Week 9, and Week 18
  Participants will complete Patient Health Questionnaire-8 to measure depression. The total score is calculated by adding up the scores of each item, and ranges from 0 to 24. The cut points for mild, moderate, moderately severe, and severe depression are 5, 10, 15, and 20, respectively.
Physical activity | Baseline, Week 9, and Week 18
  Participants will complete Physical Activity for Elderly questionnaire to measure physical activity levels. The total score is calculated using an algorithm that multiplies activity weights by activity frequencies. Higher scores correspond to greater physical activity levels.
Nutrition risk | Baseline, Week 9, and Week 18
  Participants will complete SCREEN-14 tool to measure nutrition risk. The score ranges from 0 to 64. Individuals who receive a score less than 50 are considered nutritionally at risk. A score of 2 or less from an individual response may help understand the items that put individuals at nutrition risk.
Balance | Baseline, Week 9, and Week 18
  Participants will perform a series of balance tests (side-by-side stand, semi-tandem stand, tandem stand) to assess balance. The total balance score ranges from 0 to 4 wherein the higher scores represent greater balance.
Maintenance (exercise adherence at Week 18) | Baseline, Week 9, and Week 18
  Maintenance will be reported as the adherence to the exercise sessions at the end of 18-week follow-up for immediate group only.
Quality of Life Questionnaire of the European Foundation for Osteoporosis | Baseline, Week 9, and Week 18
  Participants will complete the 41-item Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) to measure quality of life. The total score is calculated by summing each item in the questionnaire and then transforming the score to a scale from 0 to 100. Higher scores indicate a greater quality of life.
Falls | Baseline, Week 4, Week 8, and Week 16
  The number of people who fall and rate of falls will be recorded using monthly fall logs. Participants will self-report their falls.
Fear of movement | Baseline, Week 9, and Week 18
  Participants will complete Tampa Scale of Kinesiophobia to assess the participants' fear of movement related to the pain. The total score ranges from 17 to 68. The lowest score of 17 represents no or little fear of movement whereas the higher scores indicate a greater fear of movement.
Reach | At Baseline
  Reach will be reported using PROGRESS-Plus (Place; Race/ethnicity/culture/language; Occupation; Out of Work, Gender and sex; Religion, Education, Socioeconomic status, Social capital) factors to describe participants. The number of individuals recruited who are ≤12 weeks versus >12 weeks post-vertebral fracture, and those who attend outcome assessments in-person or virtually will be presented.
Adoption | Over the 5-month recruitment period
  Adoption will be reported as the number of screened and enrolled patients by referral source. The fracture verification process will also be assessed (i.e., the length of time to obtain radiology reports and number of people with ambiguous radiology reports).
Physical function | Baseline, Week 9, and Week 18
  Participants will perform the 30 Second Chair Stand Test to assess lower extremity muscle power. Scores vary depending on age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (4):
- Canada (4):
  - Arthritis Research Canada, Vancouver, British Columbia
  - Geras Centre for Aging Research, Hamilton, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Ponzano M, Tibert N, Brien S, Funnell L, Gibbs JC, Keller H, Laprade J, Morin SN, Papaioannou A, Weston ZJ, Wideman TH, Giangregorio LM. Development, Acceptability, and Usability of a Virtual Intervention for Vertebral Fractures. Phys Ther. 2023 Dec 6;103(12):pzad098. doi: 10.1093/ptj/pzad098. PMID 37555708
- [Derived] Sevinc A, Papaioannou A, Morin SN, Watt JA, Kherani RB, Brien S, Funnell L, Thabane L, Beaupre LA, Gibbs JC, Keller H, McArthur C, Ponzano M, Singh S, Straus S, Thain J, Weston ZJ, Wideman TH, Witiw CD, Giangregorio L. Virtual Intervention for Vertebral frActures (VIVA): protocol for a feasibility study of a multicentre randomized controlled trial. Pilot Feasibility Stud. 2025 Jul 5;11(1):94. doi: 10.1186/s40814-025-01665-x. PMID 40618179